CLINICAL TRIAL: NCT07242872
Title: Association Between Smartphone Addiction and Postoperative Pain and Analgesic Consumption in Adult Patients Undergoing Elective Rhinoplasty: A Prospective Observational Study
Brief Title: Screen Addiction and Postoperative Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-374
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: Smartphone; Behavior, Addictive; Analgesics; Rhinoplasty; Pain Measurement
MeSH Terms: conditions — Pain, Postoperative; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective rhinoplasty: This cohort includes adult patients aged 18-45 years with ASA physical status I-II who are scheduled to undergo elective rhinoplasty under general anesthesia. All participants will complete preoperative assessments, including demographic data and validated Turkish versions of the Smartphone Application-Based Addiction Scale and the Nomophobia Questionnaire (NMP-Q). Postoperative pain scores (VAS) will be recorded at 1, 6, 12, and 24 hours following surgery, along with total analgesic consumption within the first 24 hours. No interventions will be applied as part of the study; the cohort will be observed prospectively

SUMMARY:
Excessive or problematic smartphone use has become increasingly common and has been associated with various psychological and physical health consequences, including anxiety, depressive symptoms, reduced sleep quality, musculoskeletal pain, and heightened pain perception. Postoperative pain is influenced not only by surgical trauma but also by individual psychological and behavioral characteristics. This prospective observational study aims to investigate whether smartphone addiction levels influence postoperative pain scores and analgesic consumption in patients undergoing elective rhinoplasty surgery.

DETAILED DESCRIPTION:
Problematic smartphone use-often referred to as smartphone addiction-has emerged as a significant behavioral concern worldwide. Prior research has demonstrated associations between excessive smartphone use and anxiety, depression, sleep disturbances, impaired attention, and increased musculoskeletal discomfort. Moreover, psychological factors such as stress, anxiety, and cognitive attention patterns are known to modulate postoperative pain perception.

Individuals with higher levels of smartphone addiction commonly exhibit elevated anxiety, restlessness, and depressive symptoms, which may heighten pain sensitivity and interfere with postoperative pain coping mechanisms. However, current literature includes limited evidence directly examining the relationship between smartphone addiction and postoperative pain outcomes.

This single-center prospective observational study will include adult patients aged 18-45 years undergoing elective rhinoplasty surgery under general anesthesia. Eligible participants will be ASA physical status I-II and without psychiatric disorders, chronic analgesic or psychotropic medication use, communication difficulties, prior rhinoplasty surgery, or additional concurrent surgical procedures.

Preoperative data collection will include demographic variables (age, sex, education level, duration of daily smartphone use). Participants will complete two validated instruments in Turkish: The Smartphone Application-Based Addiction Scale - Turkish Version, The Nomophobia Questionnaire (NMP-Q) - Turkish Version.

Surgical and anesthesia management will follow standardized institutional protocols. Postoperative pain will be assessed using the Visual Analog Scale (VAS) at 1, 6, 12, and 24 hours following surgery. Total analgesic consumption within the first 24 hours will also be recorded.

Participants will be categorized based on their smartphone addiction scores, and postoperative pain outcomes and analgesic consumption will be compared between groups. Additionally, correlation analyses will be performed to explore the association between smartphone addiction levels and perceived postoperative pain.

Sample size was calculated using an effect size derived from a previous study reporting a correlation coefficient of rho = 0.292 between problematic phone use and perceived pain. With a significance level of 0.05 and a statistical power of 80%, a minimum of 91 participants were required. To compensate for an anticipated dropout rate of approximately 10%, the final planned sample size is 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years
* Scheduled for elective primary rhinoplasty under general anesthesia
* ASA physical status I-II
* Ability to provide informed consent

Exclusion Criteria:

* History of psychiatric disorders (diagnosed anxiety, depression, bipolar disorder, psychosis)
* Use of chronic analgesic, opioid, sedative, or psychotropic medication
* Previous rhinoplasty or combined surgeries
* Neurological disorders affecting pain perception
* Communication difficulties or inability to complete questionnaires
* Chronic pain syndromes (e.g., fibromyalgia, chronic back pain)
* Intraoperative complications requiring deviation from standard anesthesia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sample size was calculated using an effect size derived from a previous study reporting a correlation coefficient of rho = 0.292 between problematic phone use and perceived pain. With a significance level of 0.05 and a statistical power of 80%, a minimum of 91 participants were required. To compensate for an anticipated dropout rate of approximately 10%, the final planned sample size is 100 participants.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS) | 1st, 6th, 12th, and 24th postoperative hours.
  Pain intensity measured using the Visual Analog Scale (0-10)

SECONDARY OUTCOMES:
Total Analgesic Consumption | 24 hours postoperatively
  The total analgesic consumption within the first 24 postoperative hours, including tramadol administered through patient-controlled analgesia (PCA).

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study are available from the corresponding author upon reasonable request. Interested researchers may contact the corresponding author via email and provide a brief description of their intended use.
Supporting Information: Study Protocol, SAP, ICF